CLINICAL TRIAL: NCT02887846
Title: Comparing Heated Humidified High-flow Nasal Cannula Therapy and Nasal Continuous Positive Airway Pressure (nCPAP) Ventilation Methods for the Prevention of Extubation Failure in Preterm Infants Less Than 32 Weeks' Gestational Age: Randomized Clinical Trial
Brief Title: Comparing HHHFNC and nCPAP Ventilation Methods for the Prevention of Extubation Failure in Preterm Infants
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zekai Tahir Burak Women's Health Research and Education Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 11082016
Record Dates: First submitted 2016-08-15; First posted 2016-09-02 (Estimated); Last update posted 2016-09-13 (Estimated); Status verified 2016-08

CONDITIONS: Extubation Failure; Prematurity
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- group 1 (Active Comparator): Heated humidified high-flow nasal cannula therapy device for post extubation
  Interventions: Device: Heated Humidified High-Flow Nasal Cannula
- group 2 (Active Comparator): Nasal continuous positive airway pressure for post extubation
  Interventions: Device: Heated Humidified High-Flow Nasal Cannula

INTERVENTIONS:
Device: Heated Humidified High-Flow Nasal Cannula — Patients requiring mechanical ventilation for at least 6 hours on the first 7 postnatal days will be included in the study.When patients were Fi O2 < 0,40, Pa CO2 < 65 mmHg, pH> 7.20, MAP (mean airway pressure) <7 cm H2O, they will be extubated if statistically stable.Oxygen-air mixture of 4-6 l / min flow rate will be set in HHHFNC group, and pressure will be set to 5-8 cm H2O in NCPAP group. When flow is 2 l / min, FiO2 is<0.30 at 24 hours and above, free oxygen will be introduced. In NCPAP group, when pressure is 5 cm H2O and FiO2 < 0.30 at 24 hours and above, free oxygen will be introduced.
  Other Names: HHHFNC

SUMMARY:
Purpose is to show that HHHFNC method is as effective and safe as nCPAPand even more comfortable than it as non-invasive respiratory support for the prevention of extubation failure in preterm with gestational age of 26-32 weeks.

Patients requiring mechanical ventilation for at least 6 hours on the first 7 postnatal days will be included in the study.When patients were Fi O2 < 0,40, Pa CO2 < 65 mmHg, pH> 7.20, MAP (mean airway pressure) <7 cm H2O, they will be extubated if statistically stable.Oxygen-air mixture of 4-6 l / min flow rate will be set in HHHFNC group, and pressure will be set to 5-8 cm H2O in NCPAP group. When flow is 2 l / min, FiO2 is<0.30 at 24 hours and above, free oxygen will be introduced. In NCPAP group, when pressure is 5 cm H2O and FiO2 < 0.30 at 24 hours and above, free oxygen will be introduced.

DETAILED DESCRIPTION:
Purpose is to show that HHHFNC method is as effective and safe as nCPAP and even more comfortable than it as non-invasive respiratory support for the prevention of extubation failure in preterm with gestational age of 26-32 weeks.

Method

Primary Outcome Measures:

The effectiveness of HHHFNC and nCPAP techniques for the prevention of extubation failure within 7 days following the first extubation in preterms in need of mechanical ventilation within the first 7 postnatal days

Secondary Outcome Measures:

* the total duration of invasive and non-invasive respiratory support and the duration of free oxygen demand of patients
* Premature morbidities such as PDA, NEC, ROP, IVH, BPDand sepsis
* The degree of nasal trauma score and the degree of nasal mucosal injury
* FiO2 levels first before extubation and 6 hours after extubation
* The causes of reintubation such as apnea, acidosis, and increased need of FiO2
* The reintubation predisposing factors such as pneumothorax, atelectasis, PDA after extubation
* The weight change in the first 7-day period after extubation
* The two groups in terms of neurodevelopmental changes

Study design Patients requiring mechanical ventilation for at least 6 hours on the first 7 postnatal days will be included in the study. When patients were Fi O2 < 0,40, Pa CO2 < 65 mmHg, pH> 7.20, MAP (mean airway pressure) <7 cm H2O, they will be extubated if statistically stable. Oxygen-air mixture of 4-6 l / min flow rate will be set in HHHFNC group, and pressure will be set to 5-8 cm H2O in NCPAP group. When flow is 2 l / min, FiO2 is<0.30 at 24 hours and above, free oxygen will be introduced. In NCPAP group, when pressure is 5 cm H2O and FiO2 < 0.30 at 24 hours and above, free oxygen will be introduced.

Reintubation criteria is set as;

* FiO2 of ≥ 0.50 in order to keep oxygen saturation measured by pulse oximetry above 90 % and higher,
* Apnea requiring more than 6 alerts in a 24 -hour period in 6 consecutive hours or more than 1 apnea requiring positive pressure ventilation,
* Persistent acidosis; presence of pH < 7.20 and PCO2 > 65 mmHg in two different blood gases drawn with an interval of at least 30 minutes or treatment-resistant metabolic acidosis,
* Severe respiratory distress,
* Pulmonary haemorrhage and cardiopulmonary arrest.

ELIGIBILITY:
Inclusion Criteria: Preterm infants with gestational age between 26 weeks 0 days and 31 weeks 6 days will be included.

-

Exclusion Criteria: 1- Presence of major congenital anomaly, 2- Presence of neuromuscular disease, 3- Need of surgery within 7 days following the extubation 4- Consent not provided or refused

-

Ages: 1 Hour to 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2016-08; Primary Completion 2017-07 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
extubation failure | 7 day
  The effectiveness of HHHFNC and nCPAP techniques for the prevention of extubation failure within 7 days following the first extubation in preterms in need of mechanical ventilation within the first 7 postnatal days